CLINICAL TRIAL: NCT04528524
Title: Quality of Recovery After General Anesthesia for Elective Non-cardiac Surgery - Validation of the German Translation of the Quality of Recovery-15 Questionnaire
Brief Title: Validation of the German Quality of Recovery-15 Questionnaire
Status: Completed | Type: Observational
Sponsor: Marlene Fischer (Other)
Responsible Party: Sponsor-Investigator, Marlene Fischer, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Other Study IDs: PACQoR1
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Quality of Recovery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — QoR-15Dt

SUMMARY:
The Quality of Recovery 15-questionnaire (QoR-15) is used to assess postoperative quality of recovery after surgery and anesthesia from the patient's perspective. It evaluates five dimensions including pain, physical comfort, physical independence, psychological support, and emotional state. The aim of this study is to validate a German version of the QoR-15 scale (QoR-15Dt) to measure postoperative recovery in German-speaking patients.

ELIGIBILITY:
Inclusion Criteria:

* elective non-cardiac surgery
* fluency in German
* general anesthesia

Exclusion Criteria:

* postoperative intensive care unit admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective non-cardiac surgery under general anesthesia in a tertiary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
the German version of the QoR-15 questionnaire | first postoperative day
  Validity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No